CLINICAL TRIAL: NCT05216146
Title: Enhancement of Physical and Combat Preparedness of the Slovenian Armed Forces Members
Brief Title: Enhancement of Physical and Combat Preparedness of SAF Members
Acronym: EPCPSAF-2021
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Collaborators: Science and Research Centre Koper (Other)
Responsible Party: Principal Investigator, Armin Paravlic, Principal Investigator, University of Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 0120-495/2021/6
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Physical Fitness; Combat Readiness; Injury Prevention; Validation of Testing Batteries
Keywords: Slovenian Army; Physical Fitness; Combat Preparedness; Strength and Conditioning practice; Health; Injury prevention; Validation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All subjects except the main investigator will be blinded for group allocation and physical training program, including coaches (care provider), soldiers (participants) and outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Specially designed program for physical fitness enhancement
  Interventions: Other: Strength and Conditioning
- Control (Active Comparator): A regular program of physical exercise
  Interventions: Other: Strength and Conditioning

INTERVENTIONS:
Other: Strength and Conditioning — A specially designed strength and conditioning program will be delivered for a period of 6 months from the experienced strength and conditioning coaches. The program will consist of the basic aerobic and anaerobic exercises that could be practiced without additional equipment and with own body weight.
  Other Names: Strength and Conditioning programme

SUMMARY:
Regular and optimal fitness training has a positive effect on reducing risk or injury in addition to enhancing psychophysical and combat skills. On the other hand, excessive fitness training is one of the risk factors for injuries in soldiers. For this reason, it is necessary to establish a new system of the training process and regular monitoring of physical and combat readiness of the SAF with the help of scientific and professional methodology. The proposed research project will run for two years. The main goal of the project is to enhance physical and combat readiness and determine the epidemiology of injuries of members of the Slovenian Armed Forces (SAF). Within this aim, we will also run a validation study aimed to improve existing testing batteries for armed forces.

DETAILED DESCRIPTION:
The doctrine of Slovenian Armed Forces defines combat morale, which includes the readiness of the members of the Slovenian Armed Forces, as the greatest physical effort to overcome natural or artificial obstacles that must be overcome in the workplace or battle. Therefore, the military has specific requirements for military service. One of these is combat readiness, with physical fitness being the basis for action at the level of the human body and mind, for those who wish to achieve the skills that enable the exercise required for the professional soldier. From the viewpoint of the individual, no matter if he/she is a soldier or officer, he must be able to withstand the stresses and strains of various situations in the field, even in emergencies. This means that the body must adapt to a given situation, which requires extensive psychophysical preparation for a given situation. The profile of a high-class soldier must meet the criteria of a top athlete who is psychophysically healthy and at the highest level of his abilities when it is most needed. Certainly, there is a direct correlation between a soldier's health and his fitness, individual performance, and professional development. Throughout a career, unhealthy habits inhibit a soldier's development in the operational, self-developmental, and institutional areas of an Army leader's development strategy. Regular and optimal fitness training has a positive effect on reducing risk or injury in addition to enhancing psychophysical and combat skills. On the other hand, excessive fitness training is one of the risk factors for injuries in soldiers. For this reason, it is necessary to establish a new system of the training process and regular monitoring of physical and combat readiness of the SAF with the help of scientific and professional methodology. The proposed research project will run for two years. The goal of the project is to enhance physical and combat readiness and determine the epidemiology of injuries of members of the Slovenian Armed Forces (SAF). The results of the planned studies will be used in parallel to develop a mobile application that will facilitate the training process of SAF members and the transfer of knowledge to other interested entities and organizations. According to the project goals set, we will conduct several individual studies. Briefly, Study 1 will be a cross-sectional prospective study with the main aim to conduct an epidemiological screening of injuries and estimate the risk factors, addressing only the most common injuries (≥30 per year). Research 2 will be a longitudinal cross-sectional study in which we intend to validate testing batteries for the physical and combat readiness of SAF members. Research 3 will be a longitudinal intervention study in which we will compare the new strength and conditioning system with the existing system. We will sample adult subjects, i.e. officially employed members of the SAF (18-45 years of age, Study 1-3), of both genders, based on detailed inclusion and exclusion criteria for each study separately. The project will leave an extremely useful trail, such as a mobile application with a series of testing batteries aimed to determine physical and combat readiness, as well as preventive and rehabilitation practices for the most common injuries among SAF members. It should be emphasized that the project is limited to ensuring physical fitness for combat operations. For example, the project does not provide guidelines for the handling of firearms - that is, the accuracy of shooting, but the physical effort required to carry the weapon and prepare it for shooting. We believe that the new training system, supported by a mobile application, will come to life and provide SAF members with a more in-depth and better individualized approach to the training process, allowing individuals to optimally develop their physical and combative readiness, thus achieving greater visibility both domestically and internationally.

ELIGIBILITY:
Inclusion Criteria:

* Members of Slovenian Armed Forces with no acute and/or chronic neuromuscular and skeletal injuries and/or any other chronic disease or conditions.

Exclusion Criteria:

* older than 45 years of age
* acute and/or chronic neuromuscular and skeletal injuries
* the existence of any chronic disease or condition

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 856 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Army Combat Fitness Test (ACFT) | 75 minutes
  ACFT is testing battery used for the evaluation of physical and combat qualities of armed forces
Marine Corps Combat Fitness Test (MCCFT) | 4 minutes
  MCCFT is testing battery used for the evaluation of combat qualities of armed forces

SECONDARY OUTCOMES:
Injury occurrence | 5 minutes
  Injury occurrence evaluation
D2 test | 5 minutes
  Test of attention
Stroop test | 2 minutes
  The stroop is a neuro-psychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute.

CONTACTS AND LOCATIONS:
Overall Officials: Janez Paravlic, PhD, Study Director — Faculty of Sport; Armin Paravlic, PhD, Principal Investigator — Faculty of Sport and Science and Research Centre Koper
Locations (1):
- Faculty of Sport, Ljubljana, Slovenia, Slovenia

IPD SHARING:
Plan to Share IPD: No
There is no plan for such an action. However, if the principal investigator and the project sponsor allow this aiming to collaborate on other projects, we will be interested to do so.